CLINICAL TRIAL: NCT06718491
Title: Brief Digitally-Enhanced Intervention for Managing Emotional Pain and Reducing Alcohol Use During Medication for OUD
Brief Title: Brief Digitally-Enhanced Intervention for Reducing Alcohol Use During MOUD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Stephanie M Gorka, PhD, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024H0358
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Opioid Use Disorder
Keywords: Medications for Opioid Use Disorder; Heavy Alcohol Use; Ecological Momentary Assessments; Electroencephalography
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive one of two possible interventions.
Who Masked: Participant
Masking Description: Participants will be blind to the condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Managing Physical Reactions to Overwhelming Emotions (IMPROVE) (Experimental): In this arm, participants will receive the IMPROVE intervention, a clinician-delivered protocol targeting anxiety and uncertainty.
  Interventions: Behavioral: Managing Physical Reactions to Overwhelming Emotions (IMPROVE)
- Health Education Training (HET) (Active Comparator): In this arm, participants will receive a clinician-delivered protocol with a digital component, called HET. HET focuses on healthy living more broadly and does not include information about anxiety or uncertainty.
  Interventions: Behavioral: Health Education Training (HET)

INTERVENTIONS:
Behavioral: Managing Physical Reactions to Overwhelming Emotions (IMPROVE) — Participants may be randomized to IMPROVE. IMPROVE is a three session virtual intervention delivered by research clinicians and augmented by a mobile application. The treatment is designed to target and reduce distress contributing to heavy alcohol use during medication for opioid use disorder treatment.
  Arms: Managing Physical Reactions to Overwhelming Emotions (IMPROVE)
Behavioral: Health Education Training (HET) — Participants may be randomized to HET. HET is an active control intervention that is equally intensive as IMPROVE It includes three virtual sessions and a mobile application. HET is designed to target healthy lifestyle behaviors such as diet and sleep.
  Arms: Health Education Training (HET)

SUMMARY:
The goal of this clinical trial is to reduce heavy drinking and enhance medication for opioid use disorder (MOUD) outcomes in individuals receiving MOUD. The main questions it aims to answer are:

* Does the brief, digitally-enhanced, virtual psychotherapeutic intervention, called Managing Physical Reactions to Overwhelming Emotions (IMPROVE), impact daily alcohol use and MOUD adherence?
* Does the intervention change self-report and physiological responses to intolerance to uncertainty and anxiety sensitivity?

Researchers will compare IMPROVE to a control intervention (health education treatment) to see if IMPROVE impacts daily alcohol use and MOUD adherence.

Participants will:

* Complete a baseline electroencephalography (EEG) and self-report questionnaires.
* Complete three one-hour intervention sessions (IMPROVE or control) each one week a part.
* Complete a post-intervention EEG and self-report questionnaires.
* Complete five ecological momentary assessment (EMA) surveys a day for 21 days.
* Complete self-report questionnaires one-month after their last intervention session.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in outpatient medication for opioid use disorder (MOUD) program (within the past month)
* Heavy alcohol user defined using the National Institute on Alcohol Abuse and Alcoholism (NIAAA) criteria (i.e., consume 8+/15+ drinks per week [women/men] with at least two binge episodes [4/5+ drinks for women/men in a 2 hour period] in the past month)
* Elevated psychological distress defined as a total score of > 12 on the Kessler Psychological Distress Scale (K10; 0 to 40 range)
* 18 years of age or older
* Can read and comprehend English

Exclusion Criteria:

* Do not pass the informed decision-making capacity screener, suggesting cognitive impairment or an inability to provide informed consent
* Presence of a psychiatric or medical condition that would prevent them from providing informed consent or participating in the treatments (e.g., psychosis, mania, acute intoxication)
* Current comorbid moderate to severe substance use disorder other than alcohol and opioids
* Limited or no access to a smart phone that is compatible with the mobile application
* Participation in Phase One
* Possibility of being pregnant (by self-report)
* Current suicidal or homicidal intent indicating a need for immediate hospitalization or treatment as determined by clinical interviewer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Alcohol Use | Change from baseline to post-treatment (week 4)
  Changes in proportion of heavy drinking days and drinks per drinking day following the intervention.
Startle eyeblink potentiation during unpredictable threat | Change from baseline to post-treatment (week 4)
  Startle eyeblink potentiation will be collected during the No-, Predictable-, Unpredictable -Threat (NPU) startle paradigm. Startle is a cross-species index of aversive reactivity. Startle during unpredictable threat is an objective indicator of response to uncertain stress.
Self-reported Intolerance of Uncertainty | Change from baseline to post-treatment (week 4)
  The Intolerance of Uncertainty- Short Form is a gold-standard self-report assessment. Subscale scores on the measure range from 7-35 for 'prospective intolerance of uncertainty' and 5-25 for 'inhibitory intolerance of uncertainty', with higher scores indicating greater intolerance of uncertainty.
Late positive potential when viewing anxiety sensitivity evoking images | Change from baseline to post-treatment (week 4)
  The late positive potential will be collected from the emotional picture paradigm. The late positive potential captures emotional reactivity. Emotional reactivity to a battery of anxiety sensitivity-evoking images is an objective indicator of response to bodily anxiety sensations.
Self-reported Anxiety Sensitivity | Change from baseline to post-treatment (week 4)
  The Anxiety Sensitivity Index-3 scale is a gold standard self-report assessment. Scores range from 0 to 72 where higher scores indicate higher anxiety sensitivity.

SECONDARY OUTCOMES:
Medication Adherence | Change from baseline to post-treatment (week 4)
  Changes in proportion of days compliant with medication for opioid use disorder.
Distress-related alcohol use | Assessed multiple times a day for 21 days
  Participants will report their psychological distress and subsequent alcohol use behavior.
Daily alcohol craving | Assessed multiple times a day for 21 days
  Participants will report their alcohol craving throughout each day.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data, including electroencephalography (EEG), startle eyeblink, and behavior, from this project will be submitted to the National Institute of Mental Health Data Archive (NDA) at the subject level along with appropriate supporting documentation to enable efficient use of the data by the research community. We will follow instructions as discussed in the NDA Data Sharing Terms and Conditions.
Time Frame: The data will be submitted at the conclusion of the study.
URL: https://nda.nih.gov/